CLINICAL TRIAL: NCT02353325
Title: Iron Bioavailability From Salt Fortified With Ferrous Sulphate, Zinc Sulphate and Ascorbic Acid Encapsulated in a Polymer Jacket
Brief Title: Iron Bioavailability From Encapsulated Ferrous Sulphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Omnisalt
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; Iron fortification; Iron encapsulation
MeSH Terms: conditions — Iron Deficiencies | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- non-encapsulated FeSO4 (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4
  Interventions: Dietary Supplement: non-encapsulated FeSO4
- encapsulated FeSO4, before cooking (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4, added before cooking
  Interventions: Dietary Supplement: encapsulated FeSO4, before cooking
- encapsulated FeSO4, after cooking (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4, added after cooking
  Interventions: Dietary Supplement: encapsulated FeSO4, after cooking
- non-encapsulated FeSO4 + ascorbic acid (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4 and ascorbic acid
  Interventions: Dietary Supplement: non-encapsulated FeSO4 + ascorbic acid
- encapsulated FeSO4 + ascorbic acid, before cooking (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4 and ascorbic acid, added before cooking
  Interventions: Dietary Supplement: encapsulated FeSO4 + ascorbic acid, before cooking
- encapsulated FeSO4 + ascorbic acid, after cooking (Experimental): Maize porridge with salt fortified with non-encapsulated FeSO4 and ascorbic acid, added after cooking
  Interventions: Dietary Supplement: encapsulated FeSO4 + ascorbic acid, after cooking

INTERVENTIONS:
Dietary Supplement: non-encapsulated FeSO4
  Arms: non-encapsulated FeSO4
Dietary Supplement: encapsulated FeSO4, before cooking
  Arms: encapsulated FeSO4, before cooking
Dietary Supplement: encapsulated FeSO4, after cooking
  Arms: encapsulated FeSO4, after cooking
Dietary Supplement: non-encapsulated FeSO4 + ascorbic acid
  Arms: non-encapsulated FeSO4 + ascorbic acid
Dietary Supplement: encapsulated FeSO4 + ascorbic acid, before cooking
  Arms: encapsulated FeSO4 + ascorbic acid, before cooking
Dietary Supplement: encapsulated FeSO4 + ascorbic acid, after cooking
  Arms: encapsulated FeSO4 + ascorbic acid, after cooking

SUMMARY:
Salt is one of the very few regularly purchased food item in all socioeconomic classes including poor remote areas with subsistence farming. Therefore, it is a promising vehicle for fortification with micronutrients, such as iodine, iron, vitamin A, to alleviate the burden of micronutrient deficiencies. However, ensuring the bioavailability of iron and the sensory quality in fortified salt is difficult. Water-soluble iron compounds, such as ferrous sulphate FeSO4, are the most bioavailable, but they react with moisture and impurities in salt, and cause unacceptable changes in colour. Encapsulation can reduce iron-mediated colour change in fortified salt without significantly compromise bioavailability. In the present project we aim to investigate the iron bioavailability from salt fortified with FeSO4 using a new encapsulation type based on hyaluronic acid (HA) and a polymer from the eudragit family (EPO).

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years old
* Marginal iron status (ferritin < 25 ng/ml)
* Body weight < 65 kg
* Normal body Mass Index (18.5 - 25 kg/m2)
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by a pregnancy test) / intention to become pregnant
* Lactating up to 6 weeks before study initiation
* Moderate or severe anaemia (hemoglobin < 9.0 g/dL)
* Elevated C-reactive protein (> 5.0 mg/L)
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using Fe stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments or difficulties with blood sampling)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland